CLINICAL TRIAL: NCT06884358
Title: FunctiOnal caPaciTy Evaluation Using cardIopulMonary Testing and Stress echocArdiography in Anderson-Fabry Disease Patients: OPTIMA-FD Study
Brief Title: Functional Capacity in Anderson-Fabry Disease Patients
Acronym: OPTIMA-FD
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Massimo Piepoli, MD, PhD, IRCCS Policlinico S. Donato
Other Study IDs: OPTIMA-FD
Record Dates: First submitted 2025-01-27; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-01

CONDITIONS: Anderson-Fabry Disease
Keywords: Anderson-Fabry Disease; Cardiac Involvement; CMR; CPET
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Normal cardiac parameters and normal T1: AFD patients with normal cardiac parameters and normal T1.
- Normal cardiac parameters and reduced T1: AFD patients with no LVH and myocardial reduced T1 .
- LVH without LGE: Patients with LVH without LGE.
- Advanced cardiomyopathy with LVH and LGE: AFD patients with advanced cardiomyopathy with LVH and LGE.

SUMMARY:
The goal of this observational study is to observe the relation between excercise parameters - assessed by CPET - and rest/stress hemodynamic parameters - assessed by echocardiogram and CMR - in patients with a genetic diagnosis of Anderson-Fabry Disease.

Participants will undergo:

* baseline evaluation: clinical evaluation, disease staging with FASTEX and MSSI, KCCQ for quality of life assessment, resting 12-leads ECG, 6MWT, CPET-ESE and contrast-enhanced CMR;
* before 36 months from baseline: resting 12-leads ECG, 2D rest and stress echocardiogram, CPET-ESE, contrast-enhanced CMR, disease staging with FASTEX and MSSI and KCCQ for quality of life assessment;
* up to 7 years from baseline: clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a genetic diagnosis of AFD, according to current guidelines;
* Informed written consent with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care (for patients age <18 years old, written consent from a caregiver is mandatory).

Exclusion Criteria:

* eGFR <30 ml/min and other contraindications for CMR (relative controindication: patients with implantable device);
* Musculoskeletal limitation for exercise test on the cyclo ergometer;
* Pregnant or breastfeeding women;
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with a full comprehension of the written consent form.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with AFD from Italian referral centers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2031-11 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
CPET parameters- peak Vo2 | At baseline and before 36 months from baseline.
  Peak VO2 ml/Kg/min
CPET parameters- predicted peak Vo2 | At baseline and before 36 months from baseline.
  Predicted peak VO2 (%).
CPET parameters- VE/VCO2 slope | At baseline and before 36 months from baseline.
  VE/VCO2 slope
CPET parameters- oxygen pulse | At baseline and before 36 months from baseline.
  02 pulse (ml/beat)
CPET parameters- heart rate during exercise | At baseline and before 36 months from baseline.
  Heart rate reserve (beats/minute) Heart rate recovery (beat/minute) Heart rate recovery at one minute (beat/minute)
CPET parameters- presence of chronotropic incompetence, O2 pulse flattening and exercise oscillatory ventilation | At baseline and before 36 months from baseline.
  Chronotropic incompetence (yes/no) 02 pulse flattening (yes/no) exercise oscillatory ventilation (yes/no)
CPET parameters- VO2/work slope | At baseline and before 36 months from baseline.
  VO2/work slope (ml/min/watt)
Echocardiogram parameters- diastolic function at rest | At baseline and before 36 months from baseline.
  At rest E/A ratio. At rest mean E/E'. At rest left atrial reservoir function (%). At rest sPAP (mmHg).
Echocardiogram parameters- systolic function of the left and right ventricle at rest | At baseline and before 36 months from baseline.
  At rest TAPSE (mm) At rest LV ejection fraction (%) At rest LV stroke volume indexed for body mass surface (ml/mq) At rest right ventricular free wall strain (%)
Echocardiogram parameters- right ventricle-pulmonary artery coupling at rest. | At baseline and before 36 months from baseline.
  At rest TAPSE/sPAP (mm/mmHg)
Echocardiogram parameters- exertional diastolic function | At baseline and before 36 months from baseline.
  exertional E/A, exertional mean E/E' exertional TAPE/sPAP (mm/mmHg) mPAP/CO (mmHg/L/min)
CMR parameters - LV Mass and LV Max Wall Thickness | At baseline and before 36 months from baseline.
  LV mass (gr) and LV max wall thickness (mm).
CMR parameters - Systolic Function | At baseline and before 36 months from baseline.
  Stroke volume indexed to body surface (ml/m2) and left ventricular ejection fraction (%).
CMR parameters - T1 and T2 Mapping | At baseline and before 36 months from baseline.
  T1 and T2 mapping (msec).
CMR parameters - presence of late gadolinium enhancement | At baseline and before 36 months from baseline.
  late gadolinium enhancement (yes/no)
CMR parameters - ECV | At baseline and before 36 months from baseline.
  Extracellular volume (%)

SECONDARY OUTCOMES:
Incidence of Cardiovascular Events | Up to 7 years follow-up.
  Absolute number of all-cause mortality, CV death, ventricular arrhytmias (sustained and non-sustained VT and VF), bradyarrhytmias requiring permanent pacing, new-onset of atrial fibrillation/atrial flutter, myocardial infarction and stroke.

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Spedali Civili Hospital, Brescia, Brescia
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Milan
  - IRCCS Policlinico San Donato, San Donato Milanese, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Monza
  - Regina Margherita Hospital, Turin, Turin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Linhart A, Germain DP, Olivotto I, Akhtar MM, Anastasakis A, Hughes D, Namdar M, Pieroni M, Hagege A, Cecchi F, Gimeno JR, Limongelli G, Elliott P. An expert consensus document on the management of cardiovascular manifestations of Fabry disease. Eur J Heart Fail. 2020 Jul;22(7):1076-1096. doi: 10.1002/ejhf.1960. Epub 2020 Aug 14. PMID 32640076
- [Background] Reant P, Testet E, Reynaud A, Bourque C, Michaud M, Rooryck C, Goizet C, Lacombe D, de-Precigout V, Peyrou J, Cochet H, Lafitte S. Characterization of Fabry Disease cardiac involvement according to longitudinal strain, cardiometabolic exercise test, and T1 mapping. Int J Cardiovasc Imaging. 2020 Jul;36(7):1333-1342. doi: 10.1007/s10554-020-01823-7. Epub 2020 May 8. PMID 32385539
- [Background] Bierer G, Kamangar N, Balfe D, Wilcox WR, Mosenifar Z. Cardiopulmonary exercise testing in Fabry disease. Respiration. 2005 Sep-Oct;72(5):504-11. doi: 10.1159/000087675. PMID 16210890
- [Background] Lobo T, Morgan J, Bjorksten A, Nicholls K, Grigg L, Centra E, Becker G. Cardiovascular testing in Fabry disease: exercise capacity reduction, chronotropic incompetence and improved anaerobic threshold after enzyme replacement. Intern Med J. 2008 Jun;38(6):407-14. doi: 10.1111/j.1445-5994.2008.01669.x. PMID 18613897
- [Background] Ditaranto R, Leone O, Lovato L, Niro F, Cenacchi G, Papa V, Baldovini C, Ferracin M, Salamon I, Kurdi H, Parisi V, Capelli I, Pession A, Liguori R, Potena L, Seri M, Martin Suarez S, Galie N, Moon JC, Biagini E. Correlations Between Cardiac Magnetic Resonance and Myocardial Histologic Findings in Fabry Disease. JACC Cardiovasc Imaging. 2023 Dec;16(12):1629-1632. doi: 10.1016/j.jcmg.2023.06.011. Epub 2023 Aug 2. No abstract available. PMID 37542504
- [Background] Linhart A, Elliott PM. The heart in Anderson-Fabry disease and other lysosomal storage disorders. Heart. 2007 Apr;93(4):528-35. doi: 10.1136/hrt.2005.063818. No abstract available. PMID 17401074
- [Background] Pieroni M, Moon JC, Arbustini E, Barriales-Villa R, Camporeale A, Vujkovac AC, Elliott PM, Hagege A, Kuusisto J, Linhart A, Nordbeck P, Olivotto I, Pietila-Effati P, Namdar M. Cardiac Involvement in Fabry Disease: JACC Review Topic of the Week. J Am Coll Cardiol. 2021 Feb 23;77(7):922-936. doi: 10.1016/j.jacc.2020.12.024. PMID 33602475